CLINICAL TRIAL: NCT03247270
Title: Physical Fitness and Brain - Interventional Study of the Importance of Physical Fitness on Symptoms of Anxiety, Cognitive Ability and Sick Leave, in Primary Care.
Brief Title: Physical Fitness and Brain - Interventional Study
Acronym: PHYSBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dnr300-16
Record Dates: First submitted 2017-08-04; First posted 2017-08-11 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention I (Experimental): Physical exercise intervention: 12 week exercise program with low-intensity fitness training 3 times per week.
  Interventions: Behavioral: Intervention I
- Intervention II (Experimental): Physical exercise intervention:12 week exercise program with moderate to high-intensity fitness training 3 times per week
  Interventions: Behavioral: Intervention II
- Control group (No Intervention): Control group, who will have a physiotherapy session once and will be given general advice about physical activity.

INTERVENTIONS:
Behavioral: Intervention I — Low intensive physical exercise
  Arms: Intervention I
Behavioral: Intervention II — High intensive physical exercise
  Arms: Intervention II

SUMMARY:
According to the Global Burden of Disease report in 2015, anxiety disorders are among the top 10 contributors to years lived with disability worldwide. There is a need for effective treatment protocols. As cardiovascular fitness has a major impact on the brain's ability to change structurally and functionally, interventions involving physical exercise might prove positive in the treatment of persons with anxiety. Yet there are few high quality clinical studies with physical exercise as an intervention for anxiety disorders.

Aims:

1. To test a 12 week physical exercise intervention for persons treated for anxiety disorders within primary care. The exposure of interest is intensity of physical exercise; outcomes include anxiety symptom burden, cognitive ability and sick leave.
2. To gain knowledge regarding potential mechanisms by comparing serum levels of specific hormones and cytokines (characterized and associated with brain plasticity in animal models) before and after different intensities of exercise.

Implementation:

Patients will be randomized into 3 groups: 1) Intervention I: 12 week exercise program with low-intensity fitness training 3 times per week. 2) Intervention II: 12 week exercise program with moderate to high-intensity fitness training 3 times per week. 3) Control group, who will have a physiotherapy session once and will be given general advice about physical activity. At baseline, 12 weeks and 1 year data of cardiovascular fitness, anxiety symptoms, cognitive and working ability and biomarkers will be collected.

Impact:

If physical exercise positively affects anxiety disorders it would have significance, for the patients as well as for society. In addition to increased quality of life, it may decrease future marginalization and premature death among individuals suffering from anxiety disorders. Reducing medical and sick-leave costs would also liberate health care resources to be used elsewhere in an economically strained health care system.

DETAILED DESCRIPTION:
Overall objective To examine whether physical exercise reduces anxiety symptoms, improves cognition and decreases need of sick leave in patients with anxiety disorders in primary care.

Background Mental illness is the most common reason for unemployment in people of working age and this is a growing patient group in Swedish primary care today. A survey by the European Commission showed that 17% of the Swedish population had sought help over the past year for psychiatric problems. These figures are above average for European countries and are increasing. Sweden's costs for mental illness is around MSEK 70,000 annually - an increase of MSEK 20,000 over ten years - and the proportion of sick leave days due to a psychiatric diagnosis is currently 40%. Mental illness reduces quality of life substantially. For example, 18-year-olds with anxiety disorders have increased risk of future marginalization and have a two-fold increase in mortality not only due to suicide but several different death causes, emphasizing the importance of finding effective treatment strategies.

The ability of the adult brain to change both structurally and functionally is called brain plasticity. Both in humans and in animal models physical exercise has a major impact on brain plasticity. Physical exercise can increase neurogenesis and improve memory functions in rats, and circulating insulin-like growth factor I (IGF-I) can promote this effect. Brain-derived neurotrophic factor (BDNF), and vascular endothelial growth factor (VEGF) are also involved. In addition, there is evidence that physical activity modifies neuronal activity, increases the formation of synapses, and reduces inflammation markers, which may be correlated with neuroprotection.

The investigators have previously demonstrated an association between physical fitness and anxiety disorders, suggesting positive preventive benefits of physical exercise. The beneficial effects of exercise interventions have to date mainly been demonstrated in persons with depression.

The specific aims of this project are:

1. To test a 12 week physical exercise intervention for persons treated for anxiety disorders within primary care. The exposure of interest is intensity of physical exercise; outcomes include anxiety symptom burden, cognitive ability and sickness leave.
2. To gain knowledge regarding potential mechanisms by comparing serum levels of specific hormones (characterized and associated with brain plasticity in animal models) before and after different intensities of exercise.

Relationship to the research frontline In contrast to the literature on depression there are very few clinical studies on physical exercise as an intervention for anxiety. All six trials performed hitherto were identified as being at a high risk of bias. Higher quality trials are thus required. There is a need to investigate the role of intensity, volume, frequency and type of exercise on anxiety symptoms, cognitive function and working ability in people with anxiety disorders. Also, the putative mechanisms behind the potential effects on anxiety symptoms are not elucidated and deserve attention.

A novel feature of this study is the examination of different intensities of physical fitness-improving exercise in patients with anxiety disorders. This has not previously been performed and would yield valuable insight into dose-response associations between physical fitness and effects on the brain. Objective measurements of physical fitness and cognition are a great strength of the proposed study. Analyzing specific hormones and cytokines before and after the intervention, in relation to symptoms and functional data, may provide additional information about mechanistic aspects, treatment effect and prognosis. The proposed research also offers opportunities to develop effective treatment protocols to reduce the costs of sick-leave, an area of increasing interest world-wide.

In summary, the proposed study has the potential to provide novel and important contributions to existing scientific knowledge regarding how physical exercise influences anxiety, cognitive function and working ability in patients with anxiety disorders in primary care.

Work plan The study cohort will be patients diagnosed with anxiety disorders at six primary care centres in Gothenburg, Southern Bohuslän and Halland including patients with panic syndrome (F41.0), generalized anxiety (F41.1), mixed anxiety- and depression conditions (F41.2 and F41.3), as well as anxiety UNS (F41.9). Diagnoses and comorbidities will be determined by the study psychiatrist using the M.I.N.I (the Mini International Neuropsychiatric Interview, Swedish version 6.0.0d DSM-IV). Intervention and follow-ups will take place at Primary Care Rehab.

The investigators will exclude patients from the baseline who have physical difficulties in performing a physical exercise program, pathological ECG, previous psychiatric illnesses, ongoing abuse, increased risk of suicide as determined by the GP, those under 18, pregnant women and those over 65 years of age. An additional exclusion criterion will be physical activity level at baseline exceeding one exercise occasion per week. Both people with and without ongoing treatment with psychoactive medication will be included. Supportive contact for example with a health center nurse is not an exclusion criterion but persons with ongoing psychotherapy will not be included unless the participants, as well as the GP, are willing to take a break in therapy for the duration of the 12 week study.

Recruitment takes place at primary care centres and thus represents the individuals who seek help in primary care for anxiety. Potential participants are contacted by a study psychiatrist who has no healthcare provider relationship to the patient. Intervention and follow-ups will take place at Primary Care Rehab. Each individual must sign a statement of informed consent.

At baseline, 12 weeks and 1 year, the following data will be collected by the study physician:

* MINI International Neuropsychiatric Interview (Swedish version 6.0.0d DSM-IV)
* Use of psychoactive prescription drugs including dosage and duration
* Sick leave
* Blood pressure
* BMI
* Self-report questions about alcohol (AUDIT self-assessment scale), smoking and diet
* Established psychiatric self-assessment scales: Beck Anxiety Inventory (BAI), Montgomery Åsberg Depression Rating Scale (MADRAS) and the quality of life instrument EQ-5D.
* Test Design Fluency, which is part of the D-Kefs battery of tests and is well known and used by many psychologists within education and psychiatry. This is a standardized test, carried out within a few minutes that measures executive abilities such as creativity, response inhibition and cognitive flexibility.
* Objective measurements of physical fitness in the form of estimated maximal oxygen uptake capacity (VO2max) using Åstrand's submaximal bicycle test.
* Blood samples will be taken, by a nurse at the health center, to analyze the potential correlation of the following hormones/cytokines with symptoms and function data: S-IGF-I, S-BDNF, S-VEGF and high sensitivity CRP. The blood samples are stored in a separate, locked -70 freezer at c-lab Sahlgrenska. IVO has been notified of the establishment of a biobank (No 946).

Patients will be randomized into three groups: 1) Intervention I: 12 week exercise program with low-intensity fitness training 3 times per week. 2) Intervention II: 12 week exercise program with moderate to high-intensity fitness training 3 times per week. 3) Control group. The physiotherapists at Primary Care Rehab will perform the submaximal bicycle test and personally design the exercise program in the gym. The patients will have a one-to-one session with the physiotherapists on 2 occasions and afterwards several people will exercise at the same time in the gym.

A statistical power analysis has been performed by statistician Linus Schiöler. Based on other studies, an effect size of 0.5 difference between the groups is clinically relevant, which equates to a 5 point difference between the groups using the BAI scale. Standard deviations from a previous study using BAI as the outcome measurement were in the interval of 5-10. SD 9 was used in the calculations. Based on these assumptions, at least 60 patients in each of the treatment arms should be included to reach 80% power at the 5% significance level. Health-economic analyses will be performed using primary data generated within the project concerning health-related quality of life effects caused by the intervention and information about healthcare resources utilized. A health-economic model that depicts the clinical trial will be constructed and used for computing cost-utility measures. Moreover, the model will be constructed for performing extensive probabilistic sensitivity analyses.

Ethical considerations The Ethics Committee of the University of Gothenburg approved the study: PHYSBI intervention study: EPN Göteborg Dnr: 300-16. The control group will have a physiotherapy session once and will be given general advice about physical activity. There will be a possibility to individualize treatments i.e. the same intensity but different exercises to better fit the needs and preferences of different individuals. Coding and anonymization of data occur after data collection is complete.

Collaborations The principal investigator for this project Ass Prof Maria Åberg is the chair of the steering committee for Physical Fitness and Brain Epidemiological studies (PHYSBE) which is a multidisciplinary umbrella organization for several projects. Prof Kjell Torén from Occupational and Environmental Medicine provides epidemiological competence. Prof Margda Waern provides psychiatric expertise. Physiotherapist Louise Danielsson and Prof Kristian Bolin at the Department of Economics and Statistics have experience of clinical intervention studies.

The results will be published in international renowned peer-reviewed research journals.

ELIGIBILITY:
Inclusion Criteria:

* Panic syndrome (F41.0)
* Generalized anxiety (F41.1)
* Mixed anxiety- and depression conditions (F41.2 and F41.3)
* Anxiety UNS (F41.9)

Exclusion Criteria:

* Physical difficulties in performing a physical exercise program
* Pathological ECG
* Previous psychiatric illnesses
* Ongoing abuse
* Increased risk of suicide as determined by the GP
* Pregnant women
* Physical activity level at baseline exceeding one exercise occasion per week.
* Ongoing psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Anxiety symptom burden | 12 weeks after baseline
  Established psychiatric self-assessment scales: BAI
Anxiety symptom burden | 1 year after baseline
  Established psychiatric self-assessment scales: BAI
Anxiety symptom burden | 12 weeks after baseline
  Established psychiatric self-assessment scales: MADRS-S
Anxiety symptom burden | 1 year after baseline
  Established psychiatric self-assessment scales: MADRS-S
Anxiety symptom burden | 12 weeks after baseline
  Established psychiatric self-assessment scales: EQ-5D
Anxiety symptom burden | 1 year after baseline
  Established psychiatric self-assessment scales: EQ-5D
Cognitive ability | 12 weeks after baseline
  Test Design Fluency, which is part of the D-Kefs battery of tests
Cognitive ability | 1 year after baseline
  Test Design Fluency, which is part of the D-Kefs battery of tests
Cognitive ability | 12 weeks after baseline
  Digit test included in WAIS test battery
Cognitive ability | 1 year after baseline
  Digit test included in WAIS test battery
Sick leave | 12 weeks after baseline
  Questionnaire
Sick leave | 1 year after baseline
  Questionnaire
Biomarkers in serum | 12 weeks after baseline
  S-IGF-I
Biomarkers in serum | 1 year after baseline
  S-IGF-I
Biomarkers in serum | 12 weeks after baseline
  S-BDNF
Biomarkers in serum | 1 year after baseline
  S-BDNF
Biomarkers in serum | 12 weeks after baseline
  S-VEGF
Biomarkers in serum | 1 year after baseline
  S-VEGF
Biomarkers in serum | 12 weeks after baseline
  S-high sensitivity CRP
Biomarkers in serum | 1 year after baseline
  S-high sensitivity CRP
Biomarkers in serum | 12 weeks after baseline
  S-irisin
Biomarkers in serum | 1 year after baseline
  S-irisin

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Nilsson, PhD, Study Chair — Göteborg University
Locations (1):
- Department of Public Health and Community Medicine, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Love J, Hensing G, Soderberg M, Toren K, Waern M, Aberg M. Future marginalisation and mortality in young Swedish men with non-psychotic psychiatric disorders and the resilience effect of cognitive ability: a prospective, population-based study. BMJ Open. 2016 Aug 10;6(8):e010769. doi: 10.1136/bmjopen-2015-010769. PMID 27515748
- [Background] Hillman CH, Erickson KI, Kramer AF. Be smart, exercise your heart: exercise effects on brain and cognition. Nat Rev Neurosci. 2008 Jan;9(1):58-65. doi: 10.1038/nrn2298. PMID 18094706
- [Background] Aberg MA, Aberg ND, Palmer TD, Alborn AM, Carlsson-Skwirut C, Bang P, Rosengren LE, Olsson T, Gage FH, Eriksson PS. IGF-I has a direct proliferative effect in adult hippocampal progenitor cells. Mol Cell Neurosci. 2003 Sep;24(1):23-40. doi: 10.1016/s1044-7431(03)00082-4. PMID 14550766
- [Background] Carro E, Nunez A, Busiguina S, Torres-Aleman I. Circulating insulin-like growth factor I mediates effects of exercise on the brain. J Neurosci. 2000 Apr 15;20(8):2926-33. doi: 10.1523/JNEUROSCI.20-08-02926.2000. PMID 10751445
- [Background] Lee TMC, Wong ML, Lau BW, Lee JC, Yau SY, So KF. Aerobic exercise interacts with neurotrophic factors to predict cognitive functioning in adolescents. Psychoneuroendocrinology. 2014 Jan;39:214-224. doi: 10.1016/j.psyneuen.2013.09.019. Epub 2013 Sep 25. PMID 24149089
- [Background] Eliakim A, Oh Y, Cooper DM. Effect of single wrist exercise on fibroblast growth factor-2, insulin-like growth factor, and growth hormone. Am J Physiol Regul Integr Comp Physiol. 2000 Aug;279(2):R548-53. doi: 10.1152/ajpregu.2000.279.2.R548. PMID 10938244
- [Background] Kohut ML, McCann DA, Russell DW, Konopka DN, Cunnick JE, Franke WD, Castillo MC, Reighard AE, Vanderah E. Aerobic exercise, but not flexibility/resistance exercise, reduces serum IL-18, CRP, and IL-6 independent of beta-blockers, BMI, and psychosocial factors in older adults. Brain Behav Immun. 2006 May;20(3):201-9. doi: 10.1016/j.bbi.2005.12.002. Epub 2006 Feb 28. PMID 16504463
- [Background] Stranahan AM, Martin B, Maudsley S. Anti-inflammatory effects of physical activity in relationship to improved cognitive status in humans and mouse models of Alzheimer's disease. Curr Alzheimer Res. 2012 Jan;9(1):86-92. doi: 10.2174/156720512799015019. PMID 22329653
- [Background] Aberg MA, Waern M, Nyberg J, Pedersen NL, Bergh Y, Aberg ND, Nilsson M, Kuhn HG, Toren K. Cardiovascular fitness in males at age 18 and risk of serious depression in adulthood: Swedish prospective population-based study. Br J Psychiatry. 2012 Nov;201(5):352-9. doi: 10.1192/bjp.bp.111.103416. Epub 2012 Jun 14. PMID 22700083
- [Background] Aberg MA, Nyberg J, Toren K, Sorberg A, Kuhn HG, Waern M. Cardiovascular fitness in early adulthood and future suicidal behaviour in men followed for up to 42 years. Psychol Med. 2014 Mar;44(4):779-88. doi: 10.1017/S0033291713001207. Epub 2013 Jun 6. PMID 23739044
- [Background] Cooney GM, Dwan K, Greig CA, Lawlor DA, Rimer J, Waugh FR, McMurdo M, Mead GE. Exercise for depression. Cochrane Database Syst Rev. 2013 Sep 12;2013(9):CD004366. doi: 10.1002/14651858.CD004366.pub6. PMID 24026850
- [Background] Danielsson L, Papoulias I, Petersson EL, Carlsson J, Waern M. Exercise or basic body awareness therapy as add-on treatment for major depression: a controlled study. J Affect Disord. 2014 Oct;168:98-106. doi: 10.1016/j.jad.2014.06.049. Epub 2014 Jul 5. PMID 25043321
- [Background] Stubbs B, Vancampfort D, Rosenbaum S, Firth J, Cosco T, Veronese N, Salum GA, Schuch FB. An examination of the anxiolytic effects of exercise for people with anxiety and stress-related disorders: A meta-analysis. Psychiatry Res. 2017 Mar;249:102-108. doi: 10.1016/j.psychres.2016.12.020. Epub 2017 Jan 6. PMID 28088704
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Homack S, Lee D, Riccio CA. Test review: Delis-Kaplan executive function system. J Clin Exp Neuropsychol. 2005 Jul;27(5):599-609. doi: 10.1080/13803390490918444. PMID 16019636
- [Background] Åstrand P-O et al., (2003). Textbook of work physiology: physiological bases of exercise. Champaign:Human Kinetics.
- [Background] Drummond M et al., (2015). Methods for the economic evaluation of health care programmes. Oxford, United Kingdom, Oxford University Press.
- [Derived] Nyberg J, Henriksson M, Aberg ND, Wall A, Eggertsen R, Westerlund M, Danielsson L, Kuhn HG, Waern M, Aberg M. Effects of exercise on symptoms of anxiety, cognitive ability and sick leave in patients with anxiety disorders in primary care: study protocol for PHYSBI, a randomized controlled trial. BMC Psychiatry. 2019 Jun 10;19(1):172. doi: 10.1186/s12888-019-2169-5. PMID 31182054